CLINICAL TRIAL: NCT06594406
Title: The Therapeutic Effects of Combining Bifidobacterium With Creatine on Depression
Brief Title: The Effect of Oral Bifidobacterium on Exogenous Creatine Absorption in Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Yan He, Professor, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zhujiangjy-0108
Record Dates: First submitted 2024-08-06; First posted 2024-09-19 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy individuals with creatine (Experimental)
  Interventions: Dietary Supplement: Creatine
- Healthy individuals with creatine and bifidobacterium (Experimental)
  Interventions: Dietary Supplement: Bifidobacterium and creatine
- Depression individuals with placebo (Placebo Comparator): Depressed individuals with placebo and antidepressants
  Interventions: Dietary Supplement: Placebo
- Depression individuals with creatine and bifidobacterium (Experimental): Depression individuals with creatine and bifidobacterium and antidepressants
  Interventions: Dietary Supplement: Bifidobacterium and creatine

INTERVENTIONS:
Dietary Supplement: Creatine — The dosing schedule of creatine administration is 3 g daily for 4 weeks, and administration of a placebo.
  Arms: Healthy individuals with creatine
Dietary Supplement: Bifidobacterium and creatine — The dosing schedule of creatine administration is 3 g daily for 4 weeks. In parallel, the dosing schedule of bifidobacterium administration is 200 million colony-forming units (CFU) /day for 4 weeks.
  Arms: Depression individuals with creatine and bifidobacterium; Healthy individuals with creatine and bifidobacterium
Dietary Supplement: Placebo — Administration of creatine placebo and bifidobacterium placebo for 4 weeks,
  Arms: Depression individuals with placebo

SUMMARY:
The purpose of this clinical trial is to learn if Bifidobacterium has antidepressant-like effects by enhancing creatine absorption in adults. The main questions to be answered are

Does Bifidobacterium combined with creatine have better antidepressant effects? Does Bifidobacterium enhance exogenous creatine uptake?

Researchers will compare bifidobacterium combined with creatine with placebo to see if bifidobacterium combined with creatine has antidepressant effects.

Participants will:

Take bifidobacterium, creatine or placebo every day for 4 weeks. Keep a diary of their symptoms and collect blood samples.

ELIGIBILITY:
Inclusion Criteria for depression:

* Adults age 18-60 years inclusive.
* Current diagnosis of major depression disorder (MDD) identified by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (SCID-5).
* Current Hamilton Depression Scale 17 score of > 16.
* BMI (body Mass Index) between 18 and 28 kg/m²
* Right-handed

Exclusion Criteria:

* Diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder, identified by the SCID-5.
* History of or current diagnosis of acute kidney injury (AKI), chronic kidney disease (CKD) or end-stage renal disease (ESRD)
* History of seizure disorder
* Current serious suicide risk identified by the Columbia Severity Suicide Rating Scale
* Previous diagnosis of creatine deficiency syndrome or evidence of creatine deficiency syndrome
* Antibiotic use in last 30 days
* Probiotics use in last 30 days
* Positive pregnancy test
* Breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale | 4 weeks
  Comparison of Hamilton Depression Rating Scale before and after treatment

SECONDARY OUTCOMES:
Change from baseline in creatine level in blood | 4 weeks
  Comparison of creatine level in blood before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiong Cao, Doctor, Principal Investigator — Southern Medical University
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No